CLINICAL TRIAL: NCT06087120
Title: Investigate the Prognostic and Predictive Value of Circulating Tumor DNA (ctDNA) During Neoadjuvant Chemotherapy for Breast Cancer.
Brief Title: Predicting BReast cAncer Response to neoadjuVant Therapy by ctDNA Assessment
Acronym: BRAVA
Status: Recruiting | Type: Observational
Sponsor: Gene Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: GS_ZNAB
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female; Stage II Breast Cancer; Stage III Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer
Keywords: Liquid Biopsy; Circulating Tumour DNA; Vietnam; Indonesia
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The 1st samples are collected from participants of Breast cancer, phase II-III, HER2+ /or Triple Negative breast cancer will be processed and analyzed to determine detection rate of ctDNA in the blood samples before neoadjuvant chemotherapy.
  The 2nd and 3rd samples are collected from participants will be processed and analyzed to determine the change of ctDNA in the blood samples during and after neoadjuvant chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective and observational study, aiming to determine the detection rate and change of CtDNA in blood samples of cancer patients before, during and after neoadjuvant treatment.

* Determine the rate of ctDNA positivity at the time before treatment,
* Determine the rate of ctDNA positivity at the time during treatment,
* Determine the rate of ctDNA positivity at the time after neoadjuvant therapy, whether there is a change in ctDNA expression of the study population during treatment.

And aiming to investigate the relationship between ctDNA expression and MRI imaging with pCR response in neo-adjuvant therapy:

* Correlation between ctDNA detection and pCR response. Determine the percentage of Positive Prediction Value - PPV, Negative Prediction Value - NPV of ctDNA,
* Correlation between MRI imaging and pCR response. Determination of PPV, NPV of MRI
* Combination of ctDNA detection and MRI imaging in the prognosis of pCR. Determination of PPV, NPV ratio of ctDNA combined with MRI.

DETAILED DESCRIPTION:
This is a prospective and observational study recruiting Female participants aged 18 and older, who are diagnosed with stage II-III HER+/Triple Negative Breast cancer and indicated for neoadjuvant chemotherapy at University Medical Center HCMC, had FFPE sample at the time of diagnosis and operation. This study is conducted at the Medical Genetics Institute (MGI), and MRCCC Siloam Hospitals Semanggi (Indonesia) in collaboration with the University Medical Center HCMC.

Eligible neoadjuvant chemotherapy (NAC) / treatment regimen for the study:

* AC-T (Doxorubicin, Cyclophosphamid - Taxane).
* AC-TH (Doxorubicin, Cyclophosphamid - Taxane - Trastuzumab).
* TCH (Docetaxel - Carboplatin - Trastuzumab).
* TCHP (Docetaxel - Carboplatin - Trastuzumab - Pertuzumab).

Patients are allowed to change protocol if required clinically.

The potential and voluntary participants, satisfy all the inclusion/exclusion criteria will be recruited into this study.

At enrollment, each participant will answer to the pre-designed questionnaires of demographic information, medical history.

At routine visits, the participants' clinical information and routine para-clinical results such as breast ultrasound or MRI or CT scan, chest x-ray, mamography, bone or PET-CT scan, CA 15-3 will be collected by Physicians.

Participant in this study will have samples collected the following period of time.

* At enrollment (Pre-NAC, at diagnosis): 10ml of peripheral blood for ctDNA analysis and 6-8 sections of formalin-fixed paraffin-embedded (FFPE) tumor samples collected as biopsy before treatment.
* During NAC, 10ml of peripheral blood will be collected for ctDNA analysis and Ultrasound scan of neck, breast, abdomen and pelvis; chest x-ray, CA15-3; CT Scan of the neck, abdomen and pelvis (if any) will be also collected.
* Post-NAC, 10ml of peripheral blood will be collected for ctDNA analysis and Ultrasound scan of neck, breast, abdomen and pelvis; chest x-ray, CA15-3; CT Scan of the neck, abdomen and pelvis, PET-CT scan (if any) will be also collected to compare to treatment respondence between ctDNA and imaging groups.
* After surgery, 6-8 sections of formalin-fixed paraffin-embedded (FFPE) tumor samples collected.

The study end date of a participant is estimated 1 year since enrollment date.

ELIGIBILITY:
Inclusion Criteria:

* Female,18 years old and older,
* Are diagnosed with stage II-III HER2+/Triple Negative breast cancer and indicated for neoadjuvant chemotherapy,
* FFPE sample is available at the time of diagnosis and operation,
* Are voluntary to participate in the study.

Exclusion Criteria:

* Recurrent breast cancer,
* Other cancer metastasis to the breast,
* Have been or are being treated for cancer,
* Patients did not agree to participate in the studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include female, from 18 years old or above, who are diagnosed with stage II-III HER2+/Triple Negative breast cancer and indicated for neoadjuvant chemotherapy. Eligible participants will meet all of the inclusion and exclusion criteria to be recruited into this study at University Medical Center HCMC, MRCCC Siloam Hospitals Semanggi (Indonesia).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-09-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the detection rate and change of ctDNA in blood samples of cancer patients before, during, and after neoadjuvant treatment. | 12 months following up.
  * Determine the rate of ctDNA positivity at the time before treatment
  * Determine the rate of ctDNA positivity at the time during treatment
  * Determine the rate of ctDNA positivity at the time after neoadjuvant therapy whether there is a change in ctDNA expression of the study population during treatment.
To investigate the relationship between ctDNA expression and MRI imaging with pCR response in neo-adjuvant therapy. | 12 months following up.
  * Correlation between ctDNA detection and pCR response. Determine the percentage of Positive Prediction Value - PPV, Negative Prediction Value - NPV of ctDNA,
  * Correlation between MRI imaging and pCR response. Determination of PPV, NPV of MRI,
  * Combination of ctDNA detection and MRI imaging in the prognosis of pCR, Determination of PPV, NPV ratio of ctDNA combined with MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Sinh D Nguyen, PHD, Principal Investigator — MGI; Trung Q Lam, MD, Principal Investigator — University medical center HCMC; Samuel J Haryono, MD, Principal Investigator — MRCCC Siloam Hospitals Semanggi
Locations (3):
- MRCCC Siloam Hospitals Semanggi, Jakarta, Indonesia
- Vietnam (2):
  - Medical Genetics Institute, Ho Chi Minh City
  - University Medical Center HCMC, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised data with suitable study will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be share with any other person/organization than authorized in the study.
Supporting Information: Study Protocol, ICF
Time Frame: Feb 2026
Access Criteria: GS_ZNAB_ctDNA for Breast cancer

REFERENCES:
- [Background] Schneeweiss A, Mobus V, Tesch H, Hanusch C, Denkert C, Lubbe K, Huober J, Klare P, Kummel S, Untch M, Kast K, Jackisch C, Thomalla J, Ingold-Heppner B, Blohmer JU, Rezai M, Frank M, Engels K, Rhiem K, Fasching PA, Nekljudova V, von Minckwitz G, Loibl S. Intense dose-dense epirubicin, paclitaxel, cyclophosphamide versus weekly paclitaxel, liposomal doxorubicin (plus carboplatin in triple-negative breast cancer) for neoadjuvant treatment of high-risk early breast cancer (GeparOcto-GBG 84): A randomised phase III trial. Eur J Cancer. 2019 Jan;106:181-192. doi: 10.1016/j.ejca.2018.10.015. Epub 2018 Dec 5. PMID 30528802
- [Background] Gianni L, Mansutti M, Anton A, Calvo L, Bisagni G, Bermejo B, Semiglazov V, Thill M, Chacon JI, Chan A, Morales S, Alvarez I, Plazaola A, Zambetti M, Redfern AD, Dittrich C, Dent RA, Magazzu D, De Fato R, Valagussa P, Tusquets I. Comparing Neoadjuvant Nab-paclitaxel vs Paclitaxel Both Followed by Anthracycline Regimens in Women With ERBB2/HER2-Negative Breast Cancer-The Evaluating Treatment With Neoadjuvant Abraxane (ETNA) Trial: A Randomized Phase 3 Clinical Trial. JAMA Oncol. 2018 Mar 1;4(3):302-308. doi: 10.1001/jamaoncol.2017.4612. PMID 29327055
- [Background] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Background] Loibl S, O'Shaughnessy J, Untch M, Sikov WM, Rugo HS, McKee MD, Huober J, Golshan M, von Minckwitz G, Maag D, Sullivan D, Wolmark N, McIntyre K, Ponce Lorenzo JJ, Metzger Filho O, Rastogi P, Symmans WF, Liu X, Geyer CE Jr. Addition of the PARP inhibitor veliparib plus carboplatin or carboplatin alone to standard neoadjuvant chemotherapy in triple-negative breast cancer (BrighTNess): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):497-509. doi: 10.1016/S1470-2045(18)30111-6. Epub 2018 Feb 28. PMID 29501363
- [Background] Loibl S, Untch M, Burchardi N, Huober J, Sinn BV, Blohmer JU, Grischke EM, Furlanetto J, Tesch H, Hanusch C, Engels K, Rezai M, Jackisch C, Schmitt WD, von Minckwitz G, Thomalla J, Kummel S, Rautenberg B, Fasching PA, Weber K, Rhiem K, Denkert C, Schneeweiss A. A randomised phase II study investigating durvalumab in addition to an anthracycline taxane-based neoadjuvant therapy in early triple-negative breast cancer: clinical results and biomarker analysis of GeparNuevo study. Ann Oncol. 2019 Aug 1;30(8):1279-1288. doi: 10.1093/annonc/mdz158. PMID 31095287
- [Background] Gianni L, Huang CS, Egle D, Bermejo B, Zamagni C, Thill M, Anton A, Zambelli S, Bianchini G, Russo S, Ciruelos EM, Greil R, Semiglazov V, Colleoni M, Kelly C, Mariani G, Del Mastro L, Maffeis I, Valagussa P, Viale G. Pathologic complete response (pCR) to neoadjuvant treatment with or without atezolizumab in triple-negative, early high-risk and locally advanced breast cancer: NeoTRIP Michelangelo randomized study. Ann Oncol. 2022 May;33(5):534-543. doi: 10.1016/j.annonc.2022.02.004. Epub 2022 Feb 17. PMID 35182721
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Giannone G, Milani A, Geuna E, Galizia D, Biello F, Montemurro F. What is the best pharmacotherapeutic strategy for HER-2 positive breast cancer? Expert Opin Pharmacother. 2019 Jan;20(1):5-9. doi: 10.1080/14656566.2018.1543406. Epub 2018 Nov 6. No abstract available. PMID 30396301
- [Background] Montemurro F, Nuzzolese I, Ponzone R. Neoadjuvant or adjuvant chemotherapy in early breast cancer? Expert Opin Pharmacother. 2020 Jun;21(9):1071-1082. doi: 10.1080/14656566.2020.1746273. Epub 2020 Apr 1. PMID 32237920
- [Background] Stoetzer OJ, Fersching DM, Salat C, Steinkohl O, Gabka CJ, Hamann U, Braun M, Feller AM, Heinemann V, Siegele B, Nagel D, Holdenrieder S. Circulating immunogenic cell death biomarkers HMGB1 and RAGE in breast cancer patients during neoadjuvant chemotherapy. Tumour Biol. 2013 Feb;34(1):81-90. doi: 10.1007/s13277-012-0513-1. Epub 2012 Sep 15. PMID 22983919
- [Background] Bottini A, Berruti A, Tampellini M, Morrica B, Brunelli A, Gnocchi E, Brizzi MP, Aguggini S, Fara E, Alquati P, Dogliotti L. Influence of neoadjuvant chemotherapy on serum tumor markers CA 15-3, MCA, CEA, TPS and TPA in breast cancer patients with operable disease. Tumour Biol. 1997;18(5):301-10. doi: 10.1159/000218043. PMID 9276030
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Swarup V, Rajeswari MR. Circulating (cell-free) nucleic acids--a promising, non-invasive tool for early detection of several human diseases. FEBS Lett. 2007 Mar 6;581(5):795-9. doi: 10.1016/j.febslet.2007.01.051. Epub 2007 Feb 2. PMID 17289032
- [Background] Ortolan E, Appierto V, Silvestri M, Miceli R, Veneroni S, Folli S, Pruneri G, Vingiani A, Belfiore A, Cappelletti V, Vismara M, Dell'Angelo F, De Cecco L, Bianchi GV, de Braud FG, Daidone MG, Di Cosimo S. Blood-based genomics of triple-negative breast cancer progression in patients treated with neoadjuvant chemotherapy. ESMO Open. 2021 Apr;6(2):100086. doi: 10.1016/j.esmoop.2021.100086. Epub 2021 Mar 17. PMID 33743331
- [Background] Cavallone L, Aguilar-Mahecha A, Lafleur J, Brousse S, Aldamry M, Roseshter T, Lan C, Alirezaie N, Bareke E, Majewski J, Ferrario C, Hassan S, Discepola F, Seguin C, Mihalcioiu C, Marcus EA, Robidoux A, Roy JA, Pelmus M, Basik M. Prognostic and predictive value of circulating tumor DNA during neoadjuvant chemotherapy for triple negative breast cancer. Sci Rep. 2020 Sep 7;10(1):14704. doi: 10.1038/s41598-020-71236-y. PMID 32895401
- [Background] Cailleux F, Agostinetto E, Lambertini M, Rothe F, Wu HT, Balcioglu M, Kalashnikova E, Vincent D, Viglietti G, Gombos A, Papagiannis A, Veys I, Awada A, Sethi H, Aleshin A, Larsimont D, Sotiriou C, Venet D, Ignatiadis M. Circulating Tumor DNA After Neoadjuvant Chemotherapy in Breast Cancer Is Associated With Disease Relapse. JCO Precis Oncol. 2022 Sep;6:e2200148. doi: 10.1200/PO.22.00148. PMID 36170624
- [Background] Magbanua MJM, Li W, Wolf DM, Yau C, Hirst GL, Swigart LB, Newitt DC, Gibbs J, Delson AL, Kalashnikova E, Aleshin A, Zimmermann B, Chien AJ, Tripathy D, Esserman L, Hylton N, van 't Veer L. Circulating tumor DNA and magnetic resonance imaging to predict neoadjuvant chemotherapy response and recurrence risk. NPJ Breast Cancer. 2021 Mar 25;7(1):32. doi: 10.1038/s41523-021-00239-3. PMID 33767190
- [Background] Lin PH, Wang MY, Lo C, Tsai LW, Yen TC, Huang TY, Huang WC, Yang K, Chen CK, Fan SC, Kuo SH, Huang CS. Circulating Tumor DNA as a Predictive Marker of Recurrence for Patients With Stage II-III Breast Cancer Treated With Neoadjuvant Therapy. Front Oncol. 2021 Nov 12;11:736769. doi: 10.3389/fonc.2021.736769. eCollection 2021. PMID 34868925
- [Background] Magbanua MJM, Swigart LB, Wu HT, Hirst GL, Yau C, Wolf DM, Tin A, Salari R, Shchegrova S, Pawar H, Delson AL, DeMichele A, Liu MC, Chien AJ, Tripathy D, Asare S, Lin CJ, Billings P, Aleshin A, Sethi H, Louie M, Zimmermann B, Esserman LJ, van 't Veer LJ. Circulating tumor DNA in neoadjuvant-treated breast cancer reflects response and survival. Ann Oncol. 2021 Feb;32(2):229-239. doi: 10.1016/j.annonc.2020.11.007. Epub 2020 Nov 21. PMID 33232761
- [Background] Zhou Q, Gampenrieder SP, Frantal S, Rinnerthaler G, Singer CF, Egle D, Pfeiler G, Bartsch R, Wette V, Pichler A, Petru E, Dubsky PC, Bago-Horvath Z, Fesl C, Rudas M, Stahlberg A, Graf R, Weber S, Dandachi N, Filipits M, Gnant M, Balic M, Heitzer E. Persistence of ctDNA in Patients with Breast Cancer During Neoadjuvant Treatment Is a Significant Predictor of Poor Tumor Response. Clin Cancer Res. 2022 Feb 15;28(4):697-707. doi: 10.1158/1078-0432.CCR-21-3231. PMID 34862246
- See also: Health Mo: Decision No. 3128/QD-BYT on the issuance of GUIDES FOR DIAGNOSIS AND TREATMENT OF BREAST CANCER. 2020. — http://thuvienphapluat.vn/van-ban/The-thao-Y-te/Quyet-dinh-3128-QD-BYT-2020-tai-lieu-chuyen-mon-Huong-dan-chan-doan-dieu-tri-ung-thu-vu-447853.aspx